CLINICAL TRIAL: NCT03553459
Title: Hemodynamic Changes Induced by Trendelenburg Maneuver to Predict Fluid Responsiveness in Patients With Extracorporeal Membrane Oxygenation
Brief Title: Trendelenburg Maneuver Predicts Fluid Responsiveness in Patients With Extracorporeal Membrane Oxygenation (TEMPLE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEMPLE
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: fluid responsiveness; trendelenburg; extracorporeal membrane oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trendelenburg Maneuver (Experimental): Trendelenburg maneuver is performed to predict fluid responsiveness. Responders are defined by an increase in stroke volume over 15% after infusion of 500ml of crystalloid solution.
  Interventions: Diagnostic Test: Trendelenburg Maneuver

INTERVENTIONS:
Diagnostic Test: Trendelenburg Maneuver — In the Trendelenburg position, the body is laid supine, or flat on the back with the feet higher than the head by 15-30 degrees. The venous return increases in the trendelenburg position which in turn increases the stroke volume.

SUMMARY:
The purpose of the study is to verify the efficacy of using trendelenburg maneuver to predict fluid responsiveness in patients with extracorporeal membrane oxygenation

ELIGIBILITY:
Inclusion Criteria:

* patients with ECMO and mechanical ventilator support
* hypotension (MAP<65mmHg)
* required volume expansion by clinical judgement of the intensivists

Exclusion Criteria:

* severe hypotension with high dose of vasopressors
* severe valve regurgitation
* cardiac arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
responders | within 1 minute after volume expansion
  responders are defined by stroke volume increases over 15% after volume expansion of 500ml crystalloid
nonresponders | within 1 minute after volume expansion
  nonresponders are defined by stroke volume increases less than 15% after volume expansion of 500ml crystalloid

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Doctor, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China

REFERENCES:
- [Derived] Luo JC, Su Y, Dong LL, Hou JY, Li X, Zhang Y, Ma GG, Zheng JL, Hao GW, Wang H, Zhang YJ, Luo Z, Tu GW. Trendelenburg maneuver predicts fluid responsiveness in patients on veno-arterial extracorporeal membrane oxygenation. Ann Intensive Care. 2021 Jan 26;11(1):16. doi: 10.1186/s13613-021-00811-x. PMID 33496906